CLINICAL TRIAL: NCT05572333
Title: A Randomised, Double-blind, Placebo-controlled Study to Investigate the Safety and Tolerability of EP395 in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Clinical Trial to Investigate the Safety and Tolerability of EP395 in Patients With COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EpiEndo Pharmaceuticals (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EP395-003
Record Dates: First submitted 2022-09-30; First posted 2022-10-07 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: The study is double-blind, placebo-controlled and parallel-group in design.
Who Masked: Participant, Investigator
Masking Description: During the study, study participants, investigators, the sponsor, and all other persons involved in the conduct of the study will be blinded to treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EP395 (Experimental): EP395 in repeated doses. Oral, once-daily administration of 3 EP395 capsules for 12 weeks.
  Interventions: Drug: EP395
- Placebo (Placebo Comparator): Matched placebo capsule. Oral, once-daily administration of 3 placebo capsules for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EP395 — Capsule for oral use
  Arms: EP395
Drug: Placebo — Capsule for oral use
  Arms: Placebo

SUMMARY:
The aim of this clinical trial is to investigate the safety and tolerability of oral, once-daily EP395 administration in COPD patients for 12 weeks.

DETAILED DESCRIPTION:
This is a randomised, double-blind, placebo-controlled, multicentre study to assess the safety and tolerability of EP395 in COPD patients.

In this study, EP395 will be administered to COPD patients for the first time. Patients will receive either EP395 or placebo as oral capsules once-daily for 12 weeks. Safety and tolerability will be assessed, as well as effect on lung function, lung inflammation and systemic inflammation. Patients' symptoms and quality of life will be assessed with questionnaires. In a sub-set of patients, bronchoscopies will be conducted, to investigate exploratory biomarkers in bronchial brushings and bronchoalveolar lavage.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to understand the information on the nature, the scope, and the relevance of the study, and to provide voluntary, written informed consent to participate in the study before any study-related procedures
2. Men and women, aged ≥45 years
3. Women of childbearing potential must:

   1. have a negative pregnancy test (blood) at Screening and (urine) Day 1
   2. agree to use, and be able to comply with, highly effective measures of contraceptive control (failure rate less than 1% per year when used consistently and correctly) without interruption, during study participation and until 90 days after the last investigational product (IP) intake.
   3. agree to abstain from breast feeding during the study participation and for 90 days after the last IP intake.
4. Men must agree to use a condom during sexual intercourse with women of childbearing potential during treatment and for 90 days after the last IP intake and should not donate sperm during this time
5. Diagnosed with COPD for at least 2 years with FEV1/forced vital capacity (FVC) ratio <0.70 and FEV1 <70% (post bronchodilator) at Screening
6. Receiving at least one maintenance inhaled therapy (ie, long acting beta-agonist [LABA], long acting muscarinic antagonist [LAMA], LABA/LAMA, LABA/inhaled corticosteroid [ICS], LAMA/ICS, or LABA/LAMA/ICS) for at least 3 months before Screening
7. Able to tolerate the sputum induction procedure and to produce an adequate (volume and sufficient quality for cell count) sputum sample
8. Body mass index of ≥19 and ≤35 kg/m2
9. History of sputum production (bronchitic phenotype) for approximately 3 months (minimum, not consecutive) in a year
10. Up to date COVID-19 vaccination (according to local law and guidelines)

Exclusion Criteria:

1. History or presence of any clinically relevant medical condition including laboratory test abnormality or planned surgery that in the investigator's opinion could affect the patient's safety or interfere with the objectives of the study
2. Exacerbation of COPD in the 3 months before Screening
3. Change in medication for COPD in the 3 months before Screening
4. Lung function at Screening that in the investigator's opinion would indicate not safe to perform sputum induction or bronchoscopy (bronchoscopy applicable only in a subset of patients)
5. History of or active tuberculosis
6. Malignancy within the past 5 years, except removed basal cell carcinoma and resected benign colonic polyps
7. Clinically significant abnormality on 12-lead ECG including prolonged corrected QT interval by Fredericia (QTcF) (>450 msec in men or >470 msec in women; based on triplicate) at Screening and Day 1 pre-dose
8. Absolute estimated glomerular filtration rate ([eGFR cystatin C + eGFR creatinine]/2) <60mL/min according to Lund-Malmö equation at Screening
9. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 x upper limit of normal at Screening
10. Use (including prescription, over-the-counter, herbal or dietary) of cytochrome P450 (CYP) inducers within 28 days before first dosing, or strong or moderate inhibitors of CYP3A4 (including dietary eg, grapefruit juice) or P-glycoprotein (Pgp) inhibitors or oral narrow therapeutic index (TI) Pgp substrates (eg, digoxin) within 14 days before first dosing (substrates, inhibitors, and inducers are listed in https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers)
11. Use of macrolide, roflumilast, or oral corticosteroid (OCS) within 28 days before Screening
12. Ongoing antibiotic treatment at Screening
13. Use of home oxygen or home-based non-invasive ventilation 3 months before Screening
14. Use of a biological therapy within 3 months before Screening
15. Use of herbal remedies within 28 days before first dose until follow-up
16. Live vaccine within 28 days or any other vaccine within 14 days before first dose until 28 days after final dose of the IP (with the exception of COVID-19 booster and flu vaccination; see Previous and concomitant medications and therapies)
17. Positive hepatitis B surface antigen, hepatitis C antibodies, or human immunodeficiency virus 1 or 2 antibodies at Screening
18. Positive test result for severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) on Day 1
19. Positive drugs of abuse test at Screening, including cotinine only in ex-smokers for at least 3 months
20. Use of e-cigarettes and vapes
21. History of alcohol or drug misuse within 12 months before Screening
22. Pregnant and lactating women
23. Prior recovery from recent infection, including but not limited to COVID 19 within the last 30 days before first dosing with IP
24. Known hypersensitivity to macrolides or EP395 or any of the excipients (dicalcium phosphate, croscarmellose sodium, magnesium stearate, microcrystalline cellulose)
25. Participation in a study of an experimental drug within 5 half-lives or 3 months before Screening, whichever is longer
26. Dependent subjects of the sponsor or investigator (eg, employees, relatives)
27. Patients without the capacity to understand the nature and risks of the study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Assessment of adverse event (AE) occurrence | From Screening (Day -28 to Day -1) to Day 100
Vital signs: Systolic and diastolic blood pressure | Screening (Day -28 to Day -1), Day 1, Day 14, Day 28, Day 42, Day 56, Day 70, Day 84, Day 100
  Absolute values and changes from baseline will be summarized for all assessed time points
Vital signs: Pulse | Screening (Day -28 to Day -1), Day 1, Day 14, Day 28, Day 42, Day 56, Day 70, Day 84, Day 100
  Absolute values and changes from baseline will be summarized for all assessed time points
Vital signs: Body temperature | Screening (Day -28 to Day -1), Day 1, Day 14, Day 28, Day 42, Day 56, Day 70, Day 84, Day 100
  Absolute values and changes from baseline will be summarized for all assessed time points
Vital signs: Respiratory rate | Screening (Day -28 to Day -1), Day 1, Day 14, Day 28, Day 42, Day 56, Day 70, Day 84, Day 100
  Absolute values and changes from baseline will be summarized for all assessed time points
Assessment of laboratory values (haematology) | Screening (Day -28 to Day -1), Day 1, Day 14, Day 28, Day 42, Day 56, Day 70, Day 84, Day 100
  Mean corpuscular haemoglobin, mean corpuscular haemoglobin concentration, mean corpuscular volume, haematocrit, haemoglobin, platelet count, white blood cell count with differentials (neutrophils, lymphocytes, monocytes, eosinophils, basophils).
  Absolute values and changes from baseline will be summarized for all assessed time points.
Assessment of blood coagulation | Screening (Day -28 to Day -1), Day 1, Day 14, Day 28, Day 42, Day 56, Day 70, Day 84, Day 100
  International normalized ratio, prothrombin time (quick test), and activated partial thromboplastin time will be assessed.
  Absolute values and changes from baseline will be summarized for all assessed time points.
Assessment of laboratory values (biochemistry) | Screening (Day -28 to Day -1), Day 1, Day 14, Day 28, Day 42, Day 56, Day 70, Day 84, Day 100
  Liver function parameters and fasting lipids (at Screening and Day 84) will be assessed in addition to the following other parameters: bicarbonate, calcium, creatinine, creatine phosphokinase, cystatin C (screening only), fasting glucose (at Screening only), sodium, urea, estimated glomerular filtration rate (at Screening only)
  Absolute values and changes from baseline will be summarized for all assessed time points
Urinalysis | Screening (Day -28 to Day -1), Day 1, Day 28, Day 56, Day 84, Day 100
  pH, glucose, protein, blood (hemoglobin), leukocytes, ketones and nitrite will be assessed.
  Clinical abnormalities will be evaluated
ECG heart rate | Screening (Day -28 to Day -1), Day 1, Day 14, Day 28, Day 56, Day 84, Day 100
  Absolute values and changes from baseline will be summarized for all assessed time points
ECG RR interval | Screening (Day -28 to Day -1), Day 1, Day 14, Day 28, Day 56, Day 84, Day 100
  Absolute values and changes from baseline will be summarized for all assessed time points
ECG PR interval | Screening (Day -28 to Day -1), Day 1, Day 14, Day 28, Day 56, Day 84, Day 100
  Absolute values and changes from baseline will be summarized for all assessed time points
ECG QRS duration | Screening (Day -28 to Day -1), Day 1, Day 14, Day 28, Day 56, Day 84, Day 100
  Absolute values and changes from baseline will be summarized for all assessed time points
ECG QT interval (uncorrected) | Screening (Day -28 to Day -1), Day 1, Day 14, Day 28, Day 56, Day 84, Day 100
  Absolute values and changes from baseline will be summarized for all assessed time points
ECG QTcF intervals | Screening (Day -28 to Day -1), Day 1, Day 14, Day 28, Day 56, Day 84, Day 100
  Absolute values and changes from baseline will be summarized for all assessed time points
Standard routine physical examination | Screening (Day -28 to Day -1), Day 1, Day 28, Day 56, Day 84, Day 100
  A standard routine physical body examination will be performed and abnormal physical examination results will be evaluated. Clinically significant abnormalities will be reported as AEs.

SECONDARY OUTCOMES:
Sputum cells (total and differential) and inflammatory mediators | Screening (Day -28 to Day -1), Day 1, Day 42, Day 70, Day 84
  Assessment of inflammatory mediators will include mediators including interleukin (IL) 8, tumour necrosis factor (TNF)-α, IL-6, IL 1β, macrophage inflammatory protein (MIP) 1α, MIP-1β, monocyte chemotactic protein (MCP)-1, surfactant protein D (SP-D), granulocyte macrophage colony-stimulating factor (GM-CSF), IL-23, IL-33, IL-25, IL-10, neutrophil elastase (NE), matrix metalloproteinase (MMP)-9, CXC motif chemokine ligand (CXCL)1, myeloperoxidase (MPO)
Blood inflammatory markers | Day 1, Day 42, Day 84
  Including assessment of fibrinogen (FBG), C-reactive protein (CRP), TNF-α, IL-6 and α2 macroglobulin
Forced expiratory volume in 1 second (FEV1) | Screening (Day -28 to Day -1), Day 1, Day 28, Day 56, Day 84
Plasma levels of EP395 | Day 14, Day 28, Day 42, Day 56, Day 70, Day 80, Day 84
St George's respiratory questionnaire (SGRQ) | Screening (Day -28 to Day -1), Day 1, Day 28, Day 56, Day 84
Exacerbations of COPD tool (EXACT) respiratory symptoms (E-RS) | Screening (Day -28 to Day -1), daily from Day 1 to Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Sukh Dave Singh, Prof., Principal Investigator — Medicines Evaluation Unit Ltd. (MEU), Manchester, United Kingdom
Locations (6):
- Germany (3):
  - IKF Pneumologie GmbH & Co. KG, Frankfurt
  - Pneumologisches Forschungsinstitut an der LungenClinic Grosshansdorf GmbH, Großhansdorf
  - IKF Pneumologie GmbH & Co. KG Institut für klinische Forschung Pneumologie, Mainz
- United Kingdom (3):
  - Bradford Royal Infirmary, Clinical Research Facility, Bradford
  - Medicines Evaluation Unit Ltd. (MEU), Manchester
  - Southampton University Faculty of Medicine, Southampton

IPD SHARING:
Plan to Share IPD: No